CLINICAL TRIAL: NCT06573424
Title: Efficacy AND Multiomic Molecular Characterization of Tirellizumab Combined With Anlotinib in in MSS/pMMR Metastatic Colorectal Cancer: Data From a Retrospective Multicenter Study
Brief Title: Tirellizumab+Anlotinib VS Anlotinib for MSS-type CRC
Status: Completed | Type: Observational
Sponsor: fan li (Other)
Responsible Party: Sponsor-Investigator, fan li, Prof, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Other Study IDs: TKI+ICIs vs TKI
Record Dates: First submitted 2024-08-15; First posted 2024-08-27 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Colon Cancer; Immunotherapy
Keywords: Immunotherapy; Multi-omics analysis; tirellizumab; anlotinib
MeSH Terms: conditions — Colonic Neoplasms | interventions — anlotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissues were obtained from patients prior to the administration of the investigational treatment and were formalin-fixed and paraffin-embedded (FFPE). The FFPE samples were subjected to WES；The other was frozen at -80℃ for the detection and analysis of TMB and tumor immune microenvironment composition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- combination group: Patients who have been treated with anlotinib + tislelizumab
  Interventions: Combination Product: Tislelizumab+anlotinib
- control group: Patients who have been treated with anlotinib monotherapy
  Interventions: Drug: anlotinib

INTERVENTIONS:
Combination Product: Tislelizumab+anlotinib — Patients who have been treated with anlotinib + tislelizumabline
  Groups: combination group
Drug: anlotinib — Patients who have been treated with anlotinib monotherapy
  Groups: control group

SUMMARY:
To compare the efficacy and safety of tirellizumab combined with anlotinib in the treatment of mss colorectal cancer. To investigate the effective biomarker of anlotinib combined with tiralizumab

DETAILED DESCRIPTION:
This was a multicenter retrospective cohort study to compare the efficacy of tyrosine kinase inhibitor（TKI） combined with immune checkpoint inhibitors(ICIs) versus tyrosine kinase inhibitor alone in the treatment of advanced MSS colorectal cancer. Patients with MSS CRC who have been confirmed by pathology and have relapsed or failed multiline therapy were included in the study. Patients who had received tirellizumab plus anlotinib were considered the combination group, and those treated with anlotinib were classified as the monotherapy group. The efficacy and safety of the two regimens were compared. At the same time, Whole-exome sequencing and transcriptome sequencing were performed on the patients in the response and non-response groups of the combination group to reveal the characteristics of their microenvironment and search for biomarkers related to response.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Patients with mss colorectal cancer who have been confirmed by pathology and have relapsed or failed multiline therapy
* Patients who have been treated with anlotinib monotherapy(12 mg qd, d1-14; 21 days per cycle) or anlotinib(12 mg qd, d1-14; 21 days per cycle)+ tislelizumab(200 mg, once every 3 weeks)
* the presence of at least one measurable target lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

Exclusion Criteria:

* Patients with other malignant tumors
* Prior treatment with antirotinib, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibodies or any other antibody or drug that specifically targets T cell co-stimulation or checkpoint pathways
* Follow-up was less than 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced MSS type colorectal cancer between November 2020 and May 2023
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
PFS | 36 months
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)

SECONDARY OUTCOMES:
OS | 36 months
  the time from the beginning of treatmentto death of any cause
Multiomic molecular characterization of the response to combination immunotherapy | 36 months
  Including WES and RNA-seq analysis. using WES(Whole-exome sequencing) to analyse the differences in the mutational profiles between responders and non-responders. RNA-seq was used to reveal pathways and TME feature associated with the response to the combination therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No